CLINICAL TRIAL: NCT05153265
Title: Critical, Intervention, Assess: Using the CIA System as a Learning Tool to Assess Bleeding Risk in Regional Anesthesia.
Brief Title: The CIA Score: a Learner's Tool
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor-Med Ctr Line, Stanford University
Other Study IDs: 48095
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Anesthesia, Local
Keywords: regional anesthesia; peripheral nerve block; acute pain medicine
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residents: We plan to distribute a survey to the Stanford anesthesiology residents to determine their assessment of the bleeding risk of nerve blocks. The survey will list the most common nerve blocks and ask the resident anesthesiologists at Stanford whether the block is low/intermediate/high risk based on a scoring system of location relative to critical structures, compressibility, and whether bleeding or hematoma would be readily apparent.
  Interventions: Other: Survey
- Attending physicians: We plan to distribute a survey to the Stanford anesthesiology attending physicians to determine their assessment of the bleeding risk of several different nerve blocks. The survey will list the most common nerve blocks and ask Stanford anesthesiologists whether the block is low/intermediate/high risk based on their experience with nerve blocks.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — There will be no interventions for study participants. Participants will be asked to complete a survey.

SUMMARY:
The goal of this project is to use a previously described scoring system - the CIA system - as a teaching tool to help learners assess the bleeding risk of peripheral nerve blocks. We will teach the CIA system to residents, then they will complete a survey in which they apply the system to various peripheral nerve blocks. We hypothesize that the CIA system will allow learners to reach the same consensus about bleeding risk as expert opinions.

DETAILED DESCRIPTION:
Prior survey of Stanford and Palo Alto VA regional anesthesiologists showed diverging assessments of whether various blocks are considered superficial or deep. Investigators hope to have a simple systematic approach to "scoring" regional anesthesia procedures which can be used as a basis for discussion and comparison of regional expert's opinions.

A scoring system using three categories of consideration to classify any regional procedure is proposed. The following three categories, Critical, Intervention, and Assess (CIA) can be used to analyze any procedure to determine bleeding risk. A score of 0 or 1, was given to each parameter depending on whether it was absent or present. A total score can be range from 0 to 3. From this, the risk can be categorized based on the total score as low-risk (0), intermediate-risk (1) or high-risk (2 or 3).

ELIGIBILITY:
Inclusion Criteria:

* Regional Anesthesiologist and interested staff from Stanford

Exclusion Criteria:

* Non-regional anesthesiologists and non-interested staff at Stanford

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stanford Regional Anesthesia attending physicians and residents
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
CIA score by trainees | 2 months
  The bleeding risk of each peripheral nerve block as assessed by trainees, using the CIA scoring system.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsui BCH, Kirkham K, Kwofie MK, Tran Q, Wong P, Chin KJ, Sondekoppam RV. Practice advisory on the bleeding risks for peripheral nerve and interfascial plane blockade: evidence review and expert consensus. Can J Anaesth. 2019 Nov;66(11):1356-1384. doi: 10.1007/s12630-019-01466-w. Epub 2019 Aug 26. PMID 31452012
- [Background] Tsui BCH. A systematic approach to scoring bleeding risk in regional anesthesia procedures. J Clin Anesth. 2018 Sep;49:69-70. doi: 10.1016/j.jclinane.2018.06.011. Epub 2018 Jun 15. No abstract available. PMID 29909204